CLINICAL TRIAL: NCT05956210
Title: SWITCH- Surgical Ward Innovation: Telemonitoring Controlled by Healthdot Evaluation of Implementation
Brief Title: Surgical Ward Innovation: Telemonitoring Controlled by Healthdot
Acronym: SWITCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Principal Investigator, Friso Schonck, Medical Docter (M.D.), Catharina Ziekenhuis Eindhoven
Other Study IDs: nWMO-2022.061
Record Dates: First submitted 2023-05-17; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Evaluation of implementation regarding Philips Healthdot as monitoring device of hospitalized patients at one surgical ward — Hospitalized patients at one surgical ward will receive a Healthdot as monitoring device which will be used as primary monitoring after 3 months of preparation with education of hospital staff, improving infrastructure and training with application, activation and interpretation

SUMMARY:
This observational clinical, single center trial is designed to evaluate the implementation of an already validated smart monitoring device, the Philips Healthdot, on one surgical ward at the Catharina hospital in Eindhoven, The Netherlands.

This study is performed during 6 months in which all patients admitted to one surgical ward will be enrolled. Implementation is established by a step-by-step approach in which the current manually performed spot check monitoring (blood pressure, oxygen saturation, respiratory rate, heart rate, temperature and pain score), with the early warning score (EWS), is continued besides smart monitoring with the Healthdot (respiratory rate, heart rate and physical activity) during the first three months (phase 1). This phase aims at optimizing the infrastructure, education of hospital staff and practice with application/ activation and interpretation of the device. Upward of 4 months, Healthdot monitoring will be the primary monitoring method and spot check monitoring is only performed additionally in case of doubt about clinical condition or requirement of additional vital parameters.

Evaluation of the implementation will be performed with a focus group and various questionnaire regarding fidelity, acceptability, adoption, feasibility, appropriateness and costs. Thereby additional analysis regarding monitoring algorithms will be performed.

DETAILED DESCRIPTION:
This project is a 6 months monocenter prospective cohort study at the Catharina hospital in the Netherlands. Every patient admitted to the one surgery department will receive a Healthdot. Implementation of the Healthdot will be performed stepwise. During phase 1 (month 1-3, the pre-implementation phase), the current standard method of care with manual spot checks and EWS will be continued. During this phase Healthdots will be applied only for training purposes in preparation to the implementation phase, phase 2 (month 3-6). This phase consists of primarily Healthdot monitoring and manual spot checks only if indicated. After these 6 months, the implementation will be evaluated and optimized and potentially extended.

Participants:

The main research population for answering the research objectives are the nurses working at the specific surgical ward at the Catharina hospital.

In total amount of 500 patients, 250 during each phase, admitted to one surgical ward at the Catharina hospital will participate and receive a Healthdot as the new standard of care. These patients will sign informed consent for use of anonymized data. This population differs in age, gender, admission cause, admission duration and comorbidities but reflects the demographics of the general population on this ward which is essential to investigate implementation and prevent selection bias.

ELIGIBILITY:
Nurses and physicians form the primary research population.

- Nurses and physicians, participating in het focus group will sign informed consent.

Patients won't be included for participation since the Healthdot will be the new standard of care regarding monitoring. Patients will however sign informed consent at admission for use of anonymized data.

Inclusion Criteria:

Nurses

* Registered in the national register of medical professions (Big register)
* Appointed as a nurse at the Catharina hospital and working at the surgical department during the study period
* Willingness to participate in the core group for evaluation of the implementation

Physicians

* Registered in the national register of medical professions (Big register)
* Appointed at the Catharina hospital as a physician or resident during the study period.
* Willingness to participate in the core group for evaluation of the implementation

Exclusion Criteria:

Nurses & Physicians

* Termination of employment within the study period
* No voluntarily participation in the core group evaluation meetings

Contra-indications for applying Healthdot

* Known to have severe allergy for the tissue adhesive used in the Healthdot.
* Any skin condition, for example prior severe rash, discoloration, scars or open wounds at the area of application
* Pregnant, or breastfeeding
* Use of topicals that are known to irritate the skin at the application area (such as medical and non-medical creams or lotions)
* Patient with active implantable device such as a Implantable Cardiac Defibrillator (ICD) or pacemaker
* Unable to understand instructions
* Left lower rib (place where Healthdot will be applied) is involved in the area of surgery, area of disinfection or area where bandages are needed.
* Transfer to a different ward during hospitalization

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The main research population for answering the research objectives are the nurses and physicians working at the specific surgical ward at the Catharina hospital. In total around 500 adult patients, 250 during each phase, admitted to one surgical ward at the Catharina hospital will participate and receive a Healthdot. These patients will sign informed consent for use of anonymized data. This population differs in age, gender, admission cause, admission duration and comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the implementation of a continuous monitoring method on the surgical ward | Conducted on a daily base during the entire study, month 1-6
  Workload: the experienced workload for nursing staff during the implementation of the Healthdot measured with the IWS and during focus group analysis

SECONDARY OUTCOMES:
Adoption | 3 focus groups sessions at month 3, 5 and 6
  The intention and attitude towards the use of the Healthdot monitoring method. Measured with evidence-based practise attitude scale (EBPAS)
Feasibility of the Healthdot | 3 focus groups sessions at month 3, 5 and 6
  The extent to which the Healthdot monitoring method can be successfully carried out by the healthcare employees. Measured with a thematic analysis and input from the core group (Braun and Clark)
Acceptability | Evaluated at month 4 and 6
  The additional effort regarding the amount of spot checks per hospital admission day per patient. Calculated with data from the electronic patient file records
Appropriateness | Evaluated after at month 4 and 6
  Relation between device false alarms (noise) and correct alarms based on the alarming protocol. Measured as signal to noise ratio (SNR)
Usability | Evaluated after at month 4 and 6
  Number of unexpected events that occur during or result from the use of the Healthdot medical device. Measured as adverse device events (ADE)
Feasibility and effectiveness | Manual time measurement during month 1-6, 2 times a week at different days
  The amount of time needed to perform and process a complete manual spot check or digital monitoring check. Measured by manual time measurement
Costs | After completing of the study at 6 months
  Cost-effectiveness analysis based on the duration of admission, the associated admission costs and the monitoring method. Calculation based on provided care and associated costs
Algorithm improvement | After completing of the study at 6 months
  Advanced algorithm analyses for improved monitoring protocols with use of artificial intelligence (AI)

CONTACTS AND LOCATIONS:
Overall Officials: Friso Schonck, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schonck F, Luyer M, van der Meer N, Bouwman A, Nienhuijs S. Implementation of a surgical ward innovation: Telemonitoring controlled by healthdot [SWITCH-trial PROTOCOL]. PLoS One. 2025 May 7;20(5):e0322472. doi: 10.1371/journal.pone.0322472. eCollection 2025. PMID 40333921

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05956210/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05956210/ICF_001.pdf